CLINICAL TRIAL: NCT06954012
Title: Effect of STRAIN COUNTER-STRAIN ON PATIENTS WITH ACUTE and POSTACUTE LATERAL ANKLE SPRAINS
Brief Title: Effect of STRAIN COUNTER-STRAIN ON PATIENTS WITH ANKLE SPRAINS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Ahliyya Amman University (Other)
Responsible Party: Principal Investigator, Atef Nadier, Assistant professor of physical therapy, Al-Ahliyya Amman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10557
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Sports Medicine Injuries
Keywords: COUNTER-STRAIN, LATERAL ANKLE SPRAINS, positional release,; effect STRAIN COUNTER-STRAIN ankle sprain
MeSH Terms: interventions — Exercise; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group a (Experimental): STRAIN COUNTER-STRAIN technique will be done plus Traditional physical therapy: ( ice application , anterior-to-posterior talar mobilization , orthoses, therapeutic exercise resistance or intensity, Stretch the gastrocnemius-soleus muscle group , partial to full weight-bearing and balance board exercises).
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- group b (Active Comparator): (Traditional physical therapy) : Ice application , anterior-to-posterior talar mobilization , orthoses, therapeutic exercise resistance or intensity, Stretch the gastrocnemius-soleus muscle group , partial to full weight-bearing balance board exercises.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION; Other: Exercise

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — ice every 2 waking hours during the first 24 to 48 hours,a brace early in rehabilitation , strain counters strain technique
Other: Exercise — RICE, anterior-to-posterior talar mobilization, orthoses
  Arms: group b

SUMMARY:
patients (male and female) will be participate at the study complain of acute to subacute ankle sprain.

Orthopedic surgeons who will be responsible for the diagnosis of the all cases. The patients will under went to anterior drawer test .

DETAILED DESCRIPTION:
Age, six, height, weight (Between 15 to 40 y).

1. FAAM TEST
2. single-leg loading (SLL) test, fOR proprioception
3. Knee to Wall Dorsiflexion Lunge Test for Ankle dorsiflexion ROM. From sitting.(MODIFIED).
4. Pain (VAS)

ELIGIBILITY:
Inclusion Criteria:

acute to subacute ankle sprain positive ankle anterior drawer test

Exclusion Criteria:

* Recurrent ankle sprain,

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
assess Pain changes | At base line and after 3months of treatment
  be visual analogue scale

SECONDARY OUTCOMES:
The Foot and Ankle Ability Measure(FAAM TEST) | At base line and after 3months of treatment
  changes of ankle function will be recorded by FAAM questionnaire
Changes of Knee to Wall Dorsiflexion Lunge Test | at base line and after 3month of treatment
  functional range of motion for ankle Dorsiflexion
changes of single-leg loading (SLL) test | at base line and after 3month of treatment
  the test assess ankle proprioception

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Al-Ahliyya Amman University, Amman
  - Hossam Metwally, Amman

IPD SHARING:
Plan to Share IPD: No